CLINICAL TRIAL: NCT01612780
Title: Trans-Nasal Maxillary Multi-Sinus Balloon Dilation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Entellus Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2233-001
Record Dates: First submitted 2012-06-01; First posted 2012-06-06 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Sinusitis
Keywords: Sinusitis; Sinus balloon dilation patients
MeSH Terms: conditions — Sinusitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- XprESS Multi-Sinus Dilation Tool (Experimental): Balloon sinus dilation
  Interventions: Device: XprESS Multi-Sinus Dilation Tool

INTERVENTIONS:
Device: XprESS Multi-Sinus Dilation Tool — Sinus balloon dilation
  Other Names: Sinus balloon dilation

SUMMARY:
The purpose of this study is to show clinically meaningful improvement in symptom severity after transnasal balloon dilation of the maxillary sinus outflow tract with or without balloon dilation of the frontal or sphenoid sinuses.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, single arm, post-approval study conducted under a common protocol designed to evaluate outcomes following trans-nasal balloon dilation of the maxillary sinus outflow tract with or without concurrent balloon dilation of the frontal or sphenoid sinuses and without any concomitant conventional sinus surgery (ie, uncinectomy, complete or partial ethmoidectomy).

ELIGIBILITY:
Inclusion Criteria:

1. Be at least age 18 years old or older.
2. Be a candidate for transnasal balloon dilation of the maxillary sinus(es) with or without balloon dilation of the frontal or sphenoid sinus(es) using XprESS consistent with the device's Indication for Use.
3. Have a sinus CT scan within 12 months of the procedure date.
4. Be able and willing to provide consent.
5. Be willing to comply with the protocol requirements.

Exclusion Criteria:

1. Have any prior maxillary sinus surgery (eg, antrostomy, uncinectomy).
2. Require any concomitant endoscopic sinus surgery (ESS) or nasal surgery (exception: turbinate reduction) at the time of the study procedure.
3. Have any nasal surgery (eg, septoplasty) or nonmaxillary sinus surgery (eg, frontal sinusotomy, sphenoidotomy, full/partial ethmoidectomy) performed within 3 months prior to enrollment.
4. Have presence of features consistent with sinus fungal disease.
5. Be allergic to nickel or barium sulfate.
6. Be currently participating in any other drug or device clinical studies excluding postapproval or marketing registry studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2012-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Entellus Medical, Plymouth, Minnesota, United States

REFERENCES:
- [Result] Gould J, Alexander I, Tomkin E, Brodner D. In-office, multisinus balloon dilation: 1-Year outcomes from a prospective, multicenter, open label trial. Am J Rhinol Allergy. 2014 Mar-Apr;28(2):156-63. doi: 10.2500/ajra.2014.28.4043. Epub 2014 Feb 14. PMID 24598043
- See also: Entellus Medical patient-facing website about sinusitis — http://www.SinusSurgeryOptions.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Balloon Sinus Dilation: Balloon sinus dilation using the XprESS Multi-Sinus Dilation Tool
Period: Overall Study
Arm/Group | Balloon Sinus Dilation
Started | 82
Completed | 76
Not Completed | 6
Not completed — Treatment not completed | 1
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Population: All enrolled participants who underwent an attempted sinus dilation procedure.
Arm/Group | Balloon Sinus Dilation
Number analyzed (Participants) | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (16.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 35
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 82
Type of sinusitis [Count of Participants; unit: Participants]
  Chronic rhinosinusitis | 73
  Recurrent acute rhinosinusitis | 9
Baseline SNOT-20 score [Mean (Standard Deviation); unit: units on a scale] — The 20-item Sino-Nasal Outcomes Test (SNOT-20) is a validated patient-reported outcome measure for assessing the presence and severity of symptoms of chronic rhinosinusitis. Symptoms on the SNOT-20 survey are each rated on a scale from 0 (no problem) to 5 (problem as bad as it can be) and the 20 symptom scores are averaged to provide a total score ranging from 0 to 5. The minimal clinically important difference in the SNOT-20 has been determined to be a reduction greater or equal to 0.8 in the total SNOT-20 score.
  units on a scale | 2.27 (0.92)

OUTCOME MEASURES:

1. Primary Outcome: Change in SNOT-20 Score
Description: The 20-item Sino-Nasal Outcomes Test (SNOT-20) is a validated patient-reported outcome measure for assessing the presence and severity of symptoms of chronic rhinosinusitis. Symptoms on the SNOT-20 survey are each rated on a scale from 0 (no problem) to 5 (problem as bad as it can be) and the 20 symptom scores are averaged to provide a total score ranging from 0 to 5. The minimal clinically important difference in the SNOT-20 has been determined to be a reduction greater or equal to 0.8 in the total SNOT-20 score.
Time Frame: Baseline and 1-year post procedure
Population: All participants who had 1 or more sinuses successfully treated with the XprESS device and both baseline and 1-year follow-up SNOT-20 scores available for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Balloon Sinus Dilation
Number analyzed (Participants) | 75
score on a scale
  Baseline | 2.3 (0.92)
  1-Year follow-up | 0.7 (0.75)
Statistical Analysis 1: Comparison: Balloon Sinus Dilation; Study sample size was established to test the hypothesis that the mean SNOT-20 score is reduced by at least 0.8 points from baseline to 1 year post procedure. Using this delta, a 1-sided alpha of 0.25, and 90% power, a sample size of 19 participants was adequate to test the hypothesis; Test type: Superiority; p < 0.0001, t-test, 2 sided — Values of p <0.05 were deemed statistically significant

2. Secondary Outcome: Revision Sinus Surgery
Description: The number of participants who require revision sinus surgery to address continuing sinus symptoms.
Time Frame: 1-year post procedure
Population: All participants with 1 or more sinuses successfully treated with the XprESS device.
Measure: Count of Participants; unit: Participants
Arm/Group | Balloon Sinus Dilation
Number analyzed (Participants) | 81
Participants | 1

3. Secondary Outcome: Number of Participants With Serious Device and/or Procedure-related Adverse Events
Description: Serious adverse events that are considered to be possibly, probably, or definitely related to the balloon device and/or dilation procedure.
Time Frame: Through 1-year post procedure follow-up
Population: All enrolled participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Balloon Sinus Dilation
Number analyzed (Participants) | 82
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were systematically collected by standardized case report forms through 1 year post procedure.
Description: All SAEs, regardless of relationship to the study device and/or procedure, were reported. The protocol only required nonserious AEs that were classified by the Investigator as device-related and/or procedure-related to be collected.
Arm/Group | Balloon Sinus Dilation
All-Cause Mortality (participants affected / at risk) | 0/82
Serious Adverse Events (participants affected / at risk) | 1/82
Other Adverse Events (participants affected / at risk) | 0/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Balloon Sinus Dilation (N=82)
Tick-borne illness (Infections and infestations) | 1 (1) — Tick-borne illness treated with intravenous antibiotics. Not related to the study device or procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less